CLINICAL TRIAL: NCT04757662
Title: A Phase IB Study to Use Tadalafil to Overcome Immunosuppression During Chemoradiotherapy for IDH-wildtype Grade III-IV Astrocytoma
Brief Title: Tadalafil to Overcome Immunosuppression During Chemoradiotherapy for IDH-wildtype Grade III-IV Astrocytoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202103257
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Grade III Astrocytoma; Grade IV Astrocytoma; Astrocytoma, Grade IV; Astrocytoma, Grade III
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tadalafil (Experimental): * Tadalafil will be given orally once daily for a total of 60 days at a weight-normalized dose as follows:
    * 10 mg/day if weight ≤63.5 kg
    * 15 mg/day if weight >63.5 kg and ≤104.3 kg
    * 20 mg/day for weight >104.3 kg
  * Standard of care fractionated radiation therapy (RT) to 60 Gy in 30 daily fractions will be administered in this study.
  * Concurrent temozolomide (TMZ) will be administered as per standard of care, i.e., continuously (Monday through Sunday) from Day 1 of RT to the last day of RT at a daily oral dose of 75 mg/m^2 at the discretion of treating medical oncologist.
  * Adjuvant therapy will administered as per standard of care. Typically, this consists of adjuvant TMZ initiated 4 to 6 weeks after completion of RT for 6 cycles at 150-200 mg/m^2 PO per day on Days 1-5 of every 28-day cycle. Tumor-treating fields or Optune device (Novocure) as per routine clinical care during adjuvant TMZ is permitted at the discretion of the treating physician.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Tadalafil is commercially available and will be purchased by the Siteman Cancer Center and distributed to participants free of charge.
  Other Names: Cialis; Adcirca

SUMMARY:
Increasing preclinical and clinical data have shown that myeloid-derived suppressor cells (MDSCs) may represent a significant driver of immunosuppression in glioblastoma (GBM, grade IV astrocytoma) and a potential mechanism of treatment resistance to chemoradiotherapy. Tadalafil, an FDA-approved drug with inexpensive cost and excellent safety profile, has been shown to effectively reduce MDSCs and restore T-cell activation in the peripheral blood and in the tumor microenvironment. The purpose of this study is to investigate the impact of targeting MDSCs in newly diagnosed IDH-wildtype grade III-IV astrocytoma by combining tadalafil with standard of care radiation therapy (RT) and temozolomide (TMZ).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of newly diagnosed supratentorial high-grade astrocytoma (WHO grade III-IV), excluding astrocytoma of brainstem and cerebellum. However, supratentorial astrocytoma with extension to the brainstem and cerebellum is allowed at discretion of the PI. Gliosarcoma or other subvariants are allowed, including the newly defined "diffuse astrocytoma, IDH-wildtype, with molecular features of glioblastoma, WHO grade IV" (Brat et al., 2018).
* Must have recovered from the effects of surgery, postoperative infection, and other complications sufficiently that they can proceed with RT and TMZ.

  -≥ 18 years of age.
* Eligible for and planning to receive standard fractionated RT of 60 Gy with concurrent TMZ.
* Karnofsky performance status ≥ 60.
* Available archival formalin-fixed paraffin-embedded (FFPE) tumor blocks.
* Adequate organ and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
  * Platelets ≥ 100,000 cells/mm3;
  * Hemoglobin > 9.0 g/dL (Note: the use of transfusion or other intervention to achieve Hgb >9.0 g/dL is acceptable);
  * Total bilirubin ≤ 1.5 upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
  * Creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min
  * If there is history of human immunodeficiency virus (HIV) infection, patients must be on effective antiretroviral therapy, and HIV viral load must be undetectable within 6 months of study enrollment.
  * If there is history of chronic hepatitis B virus (HBV) infection, patients must have either been treated or are on suppressive therapy (as indicated), and HBV viral load must be undetectable.
  * If there is history of hepatitis C virus (HCV) infection, patients must have been treated, and HCV viral load must be undetectable.
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

* Prior cranial RT or RT to the head and neck where potential field overlap may exist
* Gliomatosis, leptomeningeal, or metastatic involvement.
* High-grade glioma with known IDH mutation. IDH status could be determined by either immunohistochemistry (IDH1-R132H mutation) or sequencing (including other uncommon variants of IDH1 and IDH2 mutations) as evaluated routinely for clinical diagnosis using a CLIA-approved assay.
* Known severe hypersensitivity to tadalafil or other PDE5 inhibitors, including history of hypotension, priapism (painful erection > 4 hours duration), blindness, or hearing loss during prior treatment with tadalafil or other PDE5 inhibitors.
* Concurrent nitrate, alpha-blocker, guanylate cyclase stimulators (eg, riociguat), or cytochrome P-450 3A4 (CYP3A4) inhibitor use. CYP3A4 inhibitors include ketoconazole, itraconazole, and ritonavir.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina, angina requiring treatment with nitrates, positive cardiac stress test without evidence of subsequent effective cardiac intervention within 90 days of planned tadalafil administration
  * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous coronary angioplasty or stent within the 90 days of planned tadalafil administration
  * New York Heart Association grade II or greater congestive heart failure within 6 months
  * Serious and inadequately controlled arrhythmia
  * Hypotension (<90/50 mm Hg) or uncontrolled hypertension (>170/100 mm Hg)
  * Left ventricular outflow obstructions, such as aortic stenosis
  * Stroke within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
  * Active peptic ulcer disease.
  * End-stage renal disease (ie, on dialysis or dialysis has been recommended).
* Unilateral blindness, hereditary retinal disorder, including retinitis pigmentosa.
* Patients treated on any other therapeutic clinical protocols within 30 days prior to registration.
* Inability to undergo contrast-enhanced MRI (e.g., due to safety reasons, such as presence of a pacemaker, or severe claustrophobia).
* Pregnant or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with psychiatric illness/social situations, including alcohol or drug abuse that in the investigator's opinion will prevent administration or completion of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Relative change of MDSCs in peripheral blood | Baseline, week 6 of RT, before the start of adjuvant TMZ (approximately 4-6 weeks after the end of RT), before the 3rd cycle of adjuvant TMZ (or approximately 3 months after the end of RT if no planned 3rd cycle of adjuvant TMZ), time of progression
Frequency of adverse events as measured by CTCAE v5.0 | Baseline through 30 days after last dose of tadalafil (estimated to be 90 days)

SECONDARY OUTCOMES:
Rate of severe lymphopenia | Within 12 weeks from start of radiation therapy
  -Defined as grade 3-4 lymphopenia per CTCAE v5.0 (absolute lymphocyte count < 500)
Progression-free survival (PFS) | 12 months after completion of radiation therapy (estimated to be 14 months)
  * PFS is defined as the time from enrollment in the trial until time of disease progression or death from any cause.
  * Progression will measured per standard clinical care based on the Response Assessment in Neuro-Oncology (RANO) working group guideline
Overall survival (OS) | 12 months after completion of radiation therapy (estimated to be 14 months)
  -OS is defined as the time from enrollment in the trial until the date of death due to any cause.
Number of imaging changes on heterogeneity diffusion imaging (HDI) | Baseline and 4-6 weeks after end of radiation therapy (estimated to be 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu